CLINICAL TRIAL: NCT04069637
Title: Serum and Urine Titanium Levels in Children With Early Onset Scoliosis Treated With Growth-Sparing Instrumentation
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Scoliosis Research Society (Other)
Responsible Party: Principal Investigator, G Ying Li, Associate Professor Of Orthopaedic Surgery, University of Michigan
Other Study IDs: HUM00163421
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Early-Onset Scoliosis Deformity of Spine
Keywords: Titanium Levels

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Early onset Scoliosis: Patients with early onset scoliosis treated with growth-sparing instrumentation (TGR, MCGR, and, VEPTR).
  Interventions: Combination Product: Growth-sparing instrumentation and titanium levels
- Control group: Patients with operative fractures.

INTERVENTIONS:
Combination Product: Growth-sparing instrumentation and titanium levels — Patients with growth-sparing instrumentation as treatment for early onset scoliosis, will have their titanium (serum and urine) levels tested, to evaluated if they have elevated titanium levels compared to a control group.
  Groups: Early onset Scoliosis

SUMMARY:
The investigators are conducting research to compare serum and urine titanium levels in children with early onset scoliosis who are being treated with certain types of metal spinal rods. These rods include traditional growing rods (TGR), magnetically-controlled growing rods (MCGR), and Vertical Expandable Prosthetic Titanium Rib (VEPTR). Children with metal rods may have elevated serum and urine titanium levels. These levels may remain elevated over time. The investigators will collect serum titanium levels from children with metal rods and children without metal rods to see if there are differences in their titanium levels. The investigators will then collect a second serum titanium level from children with metal rods at least 6 months later to see if the participants titanium levels remain elevated over time. The investigators will also collect urine titanium levels from children with metal rods to see if titanium is excreted in the urine.

ELIGIBILITY:
Inclusion Criteria:

Cases: Patients with early onset scoliosis treated with traditional growing rods (TGR), magnetically controlled growing rods (MCGR), and the Vertical Expandable Prosthetic Titanium Rib (VEPTR).

Controls: Patients with operative fractures.

Exclusion Criteria:

Cases: Patients who had a previous limited spinal fusion, conversion from one type of GSI to another, TGR with stainless steel or cobalt chromium instrumentation, and indwelling implants for 6 months or less.

Controls: Patients with indwelling implants or prior implant insertion and removal.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will be patients treated by the Pediatric Orthopaedic Surgery department at Michigan Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Serum titanium levels between groups | At enrollment
  Compare serum titanium levels in patients with EOS treated with titanium alloy TGR, MCGR, and VEPTR to age-matched controls.
Serial serum titanium levels in scoliosis patients | Roughly 6 months apart
  Collect serial serum titanium levels in patients with EOS treated with TGR, MCGR, and VEPTR.
Urine titanium levels in scoliosis patients | At enrollment
  Collect urine titanium levels in patients with EOS treated with TGR, MCGR, and VEPTR.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No